CLINICAL TRIAL: NCT00522730
Title: Sepsis, Endothelial Function, and Lipids in Critically Ill Patients With Liver Failure (SELLIFA). Randomized Controlled Trial Comparing the Tolerance on Lipids and Safety of Isocaloric Parenteral Nutrition With Enteral Nutrition.
Brief Title: Safety and Tolerance on Lipids of Parenteral and Enteral Nutrition in Critically Ill Patients With Liver Failure
Acronym: SELLIFA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Pierre-François Laterre, MD, Cliniques universitaires Saint-Luc, Université Catholique de Louvain
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SELLIFA-02; B40320072194; EudraCT n°2007-002940-86
Record Dates: First submitted 2007-08-29; First posted 2007-08-30 (Estimated); Last update posted 2009-09-03 (Estimated); Status verified 2009-09

CONDITIONS: Liver Failure; Critical Illness
Keywords: Liver failure; Liver cirrhosis; Parenteral nutrition; Enteral nutrition; Lipids; Safety; Drug tolerance
MeSH Terms: conditions — Liver Failure; Critical Illness; Liver Cirrhosis; Hyperphagia | interventions — Parenteral Nutrition; Enteral Nutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Parenteral nutrition
  Interventions: Other: Parenteral nutrition
- 2 (Active Comparator): Enteral nutrition
  Interventions: Other: Enteral nutrition

INTERVENTIONS:
Other: Parenteral nutrition — Duration : 5 days
  Arms: 1
Other: Enteral nutrition — Duration : 5 days
  Arms: 2

SUMMARY:
The purpose of the study is to determine the tolerance on lipid metabolism and the safety of short-term parenteral nutrition as compared to enteral nutrition in critically ill patients with liver failure.

DETAILED DESCRIPTION:
An impaired lipid metabolism is often found in patients with liver disease and is assumed to influence the prognosis. The central role of lipid metabolism in the pathophysiology of fatty liver disease and steatohepatitis is well established. In cirrhotic patients, serum lipid levels are mostly decreased and related to the severity of liver failure; in addition, the structure and composition of lipoproteins differ from that of healthy individuals. A reduction in high-density lipoproteins has been associated with higher cytokines levels and a poorer clinical outcome in septic patients. Furthermore, the oxidative stress induced by septic complications in critically ill patients with liver failure may lead to further hepatocellular injury and activation of systemic inflammation cascade.

In this setting, the influence of nutrition on lipid metabolism may have an impact on the severity of liver failure and associated complications. Although plasma clearance and oxidation of lipids were considered to be normal in the majority of patients with cirrhosis, most previous studies only reported the effects of an oral ingestion or parenteral infusion of lipids during a few hours.

The present randomized controlled trial will be conducted in a subgroup of patients enrolled in the SELLIFA-01 prospective study (NCT00488917). The purpose of the nutritional trial is to determine the tolerance on lipid metabolism and the safety of isocaloric short-term parenteral nutrition as compared to enteral nutrition in critically ill septic and non septic patients with liver failure. The nutrition will be delivered continuously for 5 days and will provide a daily energy supply corresponding to current resting energy expenditure as determined by indirect calorimetry, with 35% of total energy requirements as lipids, 15% as proteins (maximum 1.2g/kg ideal body weight/day), and 50% as dextrose. A tight glucose control strategy will be implemented to avoid hyperglycemia.

The trial is designed to randomly assign 15 patients in each interventional group in order to detect more than 25% increase in plasma triglycerides levels with 80% statistical power for two-tailed type I error of 5%.

ELIGIBILITY:
Inclusion Criteria:

* All consecutive patients with a diagnosis of chronic liver failure;
* Planned total nutritional support;
* Adult patient aged 18 years or above, and less than 85;
* Admission to the ICU for an expected period of > 24 hours;
* Informed consent of the patient or nearest relative.

Exclusion Criteria:

* Absolute contra-indications to enteral nutrition : total mechanical ileus, persistent vomiting, high output fistulas, uncertain gastrointestinal anastomosis;
* Absolute contra-indications to parenteral nutrition : severe hypertriglyceridemia > 6 mmol/l (> 545 mg/dL), severe diabetic ketoacidosis;
* Age less than 18 years or more than 85;
* Pregnancy, including HELLP syndrome;
* Active malignancy with metastases (localized hepatocellular carcinoma is not an exclusion criteria);
* Systemic chemotherapy in the last 4 weeks (trans-arterial chemo-embolisation for localized hepatocellular carcinoma is not an exclusion criteria);
* Acquired immunodeficiency syndrome and antiretroviral therapy;
* Refusal of the patient or nearest relative.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2007-08; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Change in plasma concentration of triglycerides, total cholesterol, HDL-cholesterol, free fatty acids, apolipoproteins, lipoprotein (a) | within 5 days

SECONDARY OUTCOMES:
Incidence of hyperglycaemia | within 5 days
Alteration of liver function | within 5 and 28 days
Gastrointestinal intolerance | within 5 days
Gastrointestinal bleeding | within 5 and 28 days
Septic complications | within 5 and 28 days
Occurence of new organ dysfunction | within 5 and 28 days
Length of stay in the intensive care unit (ICU) | within 5 and 28 days
Mortality | within 5 and 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Pierre-François Laterre, MD, Study Director — Cliniques universitaires Saint-Luc- Université Catholique de Louvain; Yvan Fleury, MD, Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Locations (1):
- Departement of intensive care, Cliniques Universitaires Saint-Luc, Université Catholique de Louvain, Brussels, Belgium